CLINICAL TRIAL: NCT04938219
Title: Treatment of Intraoperative Shivering During Caesarean Section With Gloves Filled With Warm Water: a Multicentric, Randomised, Controlled Trial
Brief Title: Shivering_Basel_Baden
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-00866; qu20Buddeberg
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Shivering
Keywords: intraoperative shivering; caesarean section; neuraxial anaesthesia

STUDY DESIGN:
Intervention Model Description: Women undergoing caesarean section under neuraxial anaesthesia will be randomised into either the treatment group or control group (2 arms).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shivering Treatment Group (Experimental): Participants will be observed, and intervention will begin when a shivering score of 2 or higher is reached. The participants in the treatment group will receive one glove filled with warm water into each hand.
  Interventions: Other: Gloves filled with warm tap water
- Control Group (No Intervention): Participants in the control group will only be observed, and not given additional treatment for the shivering.

INTERVENTIONS:
Other: Gloves filled with warm tap water — The intervention in the treatment group will consist of nonsterile gloves, filled with regular tap water at a comfortable warm temperature and sealed with a plastic clip. The temperature of the water will not be measured, the investigators will take a temperature that feels comfortable in their hands
  Arms: Shivering Treatment Group

SUMMARY:
Shivering is known to occur in around 40% of women as a side effect of neuraxial anaesthesia during caesarean section.Women undergoing caesarean section under neuraxial anaesthesia are randomised into either the treatment group or control group. Women in both groups are observed during caesarean section. This study is to test a non-pharmacological and non-invasive treatment with two groups, an intervention and a control group. In the intervention group, intraoperative shivering during caesarean section is treated by placing two surgical gloves filled with warm water into the women's hands. In the control group, women will be treated with the current standard of care, which does not include specific treatment of shivering.

DETAILED DESCRIPTION:
Shivering is an involuntary, repetitive activity of skeletal muscles that often, but not exclusively, occurs as a thermoregulatory response to cold. It is associated with neuraxial anaesthesia and is therefore a commonly observed phenomenon during caesarean sections. The main cause for this is a sympathetic block of vasoconstriction in the legs, leading to cutaneous heat loss and lower core temperature. This is not always accompanied by a cold sensation, because the perceived skin temperature is increased. Out of all common side effects of neuraxial anaesthesia, shivering is perceived as the most uncomfortable and disruptive one. It can also interfere with monitoring of blood pressure, oxygen saturation and legibility of electrocardiograms. It increases the metabolic rate and oxygen consumption by up to 400%. Therefore, lactic acid and carbon dioxide production are significantly increased. Pregnant women have reduced cardiac and pulmonary reserves and may therefore have less capacity to adapt to the increased metabolic demands caused by shivering.

The incidence of shivering during caesarean section at the University Hospital Basel was determined by a previous study to be 41.0%. Studies have been conducted about pharmacological treatment options for intraoperative shivering during caesarean section. However, pharmacological treatment in pregnant and breastfeeding women is best reduced to a minimum.

This study is to test a non-pharmacological and non-invasive treatment with two groups, an intervention and a control group. In the intervention group, intraoperative shivering during caesarean section is treated by placing two surgical gloves filled with warm water into the women's hands. In the control group, women will be treated with the current standard of care, which does not include specific treatment of shivering. The warm water method has been used by doctors to reduce shivering, but the actual effects of it have never been scientifically proven. The gloves will be used as a treatment, not a prophylactic measure. Therefore, only the women who exhibit shivering during surgery will be treated.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Age older than 18 years and younger than 40 years.
* Gestational age >36 weeks
* Shivering during regional anaesthesia for caesarean section

Exclusion Criteria:

* Inability to give informed consent
* Latex allergy
* Receiving combined spinal epidural anaesthesia (CSEA)
* Secondary spinal anaesthesia for caesarean section in patients with unsatisfactory epidural labour analgesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in intensity of shivering measured on a 5-point scale | at baseline, at 2 and 5 minutes after the first assessment, and in the post-anaesthesia recovery room (approx.1 hour)ent.
  Shivering is evaluated during caesarean section 5 minutes after intervention. Shivering is graded on a scale from 0 (No shivering) to 4 (Violent muscular activity that involves the entire upper body) .The score will be recorded before the intervention and at 2 and 5 minutes after initiation of the intervention, as well as after arrival at the recovery area. Score: 0 - No shivering.
  1. - No visible muscle activity, but one or more of piloerection, peripheral vasoconstriction or peripheral cyanosis (other causes excluded).
  2. - Muscular activity in only one muscle group.
  3. - Moderate muscular activity in more than one muscle group, but not generalized shaking.
  4. - Violent muscular activity that involves the entire upper body.

SECONDARY OUTCOMES:
Change in subjective comfort levels of the patients before and after the intervention on a 11-point scale | at baseline, at 2 and 5 minutes after the first assessment, and in the post-anaesthesia recovery room (approx.1 hour)
  Change in subjective comfort level of the participant before and after the intervention on a 11-point scale (0 being very uncomfortable; 10 being very comfortable). The patient will be asked to rate their comfort level every time a shivering score is obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Bigna Buddeberg, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (2):
- Switzerland (2):
  - Kantonsspital Baden AG, Department of Anaesthesiology, Baden, Canton of Aargau
  - University Hospital Basel; Department of Anaesthesiology, Basel

IPD SHARING:
Plan to Share IPD: No
Trial and participant data will be handled with uttermost discretion and is only accessible to authorised personnel who require the data to fulfil their duties within the scope of the study. On the eCRFs and other study specific documents, participants are only identified by a unique participant number.
  Trial and participant data will be handled with uttermost discretion and is only accessible to authorised personnel who require the data to fulfil their duties within the scope of the study. On the eCRFs and other study specific documents, participants are only identified by a unique participant number.
  The participant identification list will be stored in a locked place by the sponsor-investigator. Password access to the eCRFs will only be given to the investigators directly enrolled in recruitment of participants and capturing of data.

REFERENCES:
- See also: Paper — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3591550/